CLINICAL TRIAL: NCT04540978
Title: Motor Activity and Its Barriers at the Early Phase Post-stroke.
Brief Title: Motor Activity and Its Barriers at the Early Phase Post-stroke in Acute Care Setting.
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Collaborators: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, Michal Kafri, PhD, Principal Investigator, University of Haifa
Other Study IDs: 0787-16-TLV
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Being active early after stroke prevents secondary complications, reduces hospital length of stay and improves long-term functional outcomes. Early mobilization and early rehabilitation are the means to achieve activity at the early phase post-stroke. Performance of out-of-bed activity at an acute care setting is partially dependent on the routines used in the acute care setting, however, knowledge the knowledge about associations between clinical routines and the characteristics of out-of-bed activity is limited. Also, there is limited knowledge about institutional barriers to such activity.

Accordingly, the goal of the current study is, in acute hospital inpatient setting, to: 1) characterize stroke patients' activity according to shifts (i.e. morning and evening), 2) test associations between out-of-bed activity and patients' clinical status and 3) identify barriers to activity.

The study is a prospective observational study that monitors physical activity in people after stroke while they in an acute stroke care setting, and records berries for out-of-bed activity including being in sitting or standing and walking.

Patients are included if they admitted to the hospital within 48 hours of symptom onset, passed routine initial neurologic and nursing examinations within 48 hours of admission, and have score of 5-18 on the National Institutes of Health Stroke Scale (NIHSS). Patients are excluded if they had hemorrhagic stroke, and if they have heart failure, acute coronary syndrome, unstable hemodynamics and fractures, or if they are terminally ill.

DETAILED DESCRIPTION:
Not required

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke
* Admitted to the hospital within 48 hours of symptom onset
* Passed routine initial neurologic and nursing examinations within 48 hours of admission
* Score of 5-18 on the National Institutes of Health Stroke Scale (NIHSS).

Exclusion Criteria:

* Hemorrhagic stroke
* Heart failure
* Unstable hemodynamics
* Fractures
* Terminally ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after ischemic stroke who are admitted to Neurological department, and who are having mild-moderate stroke-related symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Time in sitting according to shift (i.e. morning or evening). | Two weeks from admission or or until discharge.
  Body position is measured by activity monitor located at the lumbar spine.
Number of steps according to shift (i.e. morning or evening). | Two weeks from admission or or until discharge.
  Number of steps is recorded by activity monitor located at the lumbar spine.
Barriers for getting out of bed. | Two weeks from admission or or until discharge.
  Barriers are documented daily in a follow-up table.

SECONDARY OUTCOMES:
Longest sitting time according to shift (i.e. morning or evening). | Two weeks from admission or or until discharge.
  Body position is measured by activity monitor located at the lumbar spine.
Longest walking time according to shift (i.e. morning or evening). | Two weeks from admission or or until discharge.
  Walking time is recorded by activity monitor located at the lumbar spine.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Kafri, PhD, Principal Investigator — University of Haifa
Locations (1):
- Tel Aviv Souraski Medical Center, Neurology Department, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No